CLINICAL TRIAL: NCT03445923
Title: Can Time-lapse Parameters be Used to Predict Pregnancy of Human Embryos?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment due to Covid-19 restrictions.
Sponsor: Fertilitetscentrum AB (Other)
Responsible Party: Principal Investigator, Thorir Hardarson, Laboratory Director, Fertilitetscentrum AB
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 954-17
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphology (No Intervention): Embryos for transfer will be selected based on standard morphological evaluation.
- TLM (Active Comparator): Embryos for transfer will be selected base on standard morphological evaluation and information from time-lapse monitoring.
  Interventions: Other: Time lapse monitoring (KID Score)

INTERVENTIONS:
Other: Time lapse monitoring (KID Score) — The unique information that is obtainable from taking Pictures each 10 minutes throughout the development of the embryos will be used in the form of a special score (KID score). The score is comprised out of several key developmental parameters.
  Arms: TLM

SUMMARY:
All patients starting an IVF-treatment at the clinics, and meeting the inclusion criteria, will be offered to participate in the study. Randomization will be performed on day 5 and the patients will be allocated into either morphology only group or time-lapse group. Embryos will be cultured to day five according to the clinics own routines. All embryos in both groups will be cultured using time-lapse incubation. In the control group the embryo selection will be based only on traditional morphological evaluation and in the treatment group a time-lapse selection model (KID Score day 5) will be used to select the embryo.

DETAILED DESCRIPTION:
The aim is to study if algorithm calculated from time-lapse photography of human embryos per se can enhance the prediction of the embryo´s reproductive potential compared to embryo morphology alone.

METHODS AND MATERIAL IVF procedure Oocytes retrieved 36±1h after hCG administration will be fertilized by either standard insemination or ICSI. The morning after oocyte retrieval (day 1) zygotes will be placed into embryo time-lapse slides for culture up to the day of transfer (day 5). During the culture time, embryos will be kept in commercially available culture media and will not be removed from the time-lapse incubator until day of transfer. Embryos interact with the media and will be allowed to develop the blastocyst stage (5-6 days culture) at which time selection for transfer will be made. During the in vitro culture a single image captured in the time-lapse incubator will be used to routinely morphologically grade embryos, according to the Istanbul consensus. On day 5, developing embryos will be assessed (according to study vs. control group criteria) to select the embryo for transfer into the patient. Supernumerous GQE will be cryopreserved for future use.

Time-lapse photography All embryos will be placed in wells of time-lapse culture dishes (Embryoscope) according to the instructions of the manufacturer. Embryos in both groups will be cultured to the blastocyst stage without any media change. The time-lapse system is comprised of a desktop incubator that controls it´s environment (pH, CO2 and O2) as well as taking pictures in up to 11 focal planes for the whole duration of the culture periods.

Morphological scoring Embryo morphology will be scored according to the Gardner score and then translated to the Istanbul consensus system if needed for publication.

To assure that all embryologists annotate the embryo development correctly as well as score the blastocysts in the same way, a validation process will be performed before the onset of the study. The standardization will be accomplished through a process where the embryologists will score 20 blastocysts at day 5-development stage, which will be provided on a CD, imitating the procedure will be performed routinely in the laboratory. The embryologists will have to be approved in order to be allowed to score embryos in the study.

Embryo evaluation (both groups). Embryos will be cultured in the Embryoscope time-lapse system until day 5. If two or more blastocyst of good quality (GQB), i.e. fulfilling a minimum morphological criteria of 3BB or better, develop, a preliminary decision is made on which embryo to select for transfer. Thereafter the couple is randomized into either the control or the time-lapse group.

Decision making in the time-lapse group If the couple is randomized into the time-lapse group all embryos that have reached the blastocyst stage will be annotated. The blastocyst with the highest KID (day 5) score will be chosen for transfer. To ensure a reliable KID scores can be attained the morphological events; time to 2, 3, 4, and 5 cells, time to start of blastulation (tSB), and TE scores must be evaluated.

Decision making in the control group If the couple are randomized to the control group, the preliminary embryo selection decision will be maintained.

Study monitoring. A Data Study Monitoring Board (DSMB) Group will be assigned and have the task of conducting both safety checks and an interim analysis (planned when ca 50% of the patients have been recruited).

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing IVF or ICSI (intracytoplasmic sperm injection) that do not meet the exclusion criteria.
* The couple shall receive and sign written information about the study.
* On day 5, before the randomization the couple must have at least 2 transferrable blastocysts in order to be included in the study.

Exclusion Criteria:

* If double embryo transfer, for any reason, is planned.
* Prior participation in the study.
* Pre-implantation genetic diagnosis (PGD) treatment.
* Embryo transfer on another day than day 5.
* Oocyte cryopreservation.
* Planned total freeze of embryos for any reason (cancer, OHSS etc.)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 776 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy (week 6-7) | Patient is assessed 6-7 weeks after embryo transfer
  A confirmed pregnancy by ultrasound in the 6-7th week of gestation.

SECONDARY OUTCOMES:
Positive pregnancy tests, 18 days after embryo transfer. | Patient is assessed 2 weeks after embryo transfer by taking a pregancy test
  A pregnancy test is taken (Urine).
Early pregnancy loss (positive pregnancy test but no gestational sac observed at sonography) | Same time frame as for the primary outcome i.e. 6-7 weeks.
  This is the loss of pregnancy between positive pregnancy test (2 weeks) and ultrasound (6-7 weeks)
Correlation between the preliminary decisions of embryo fate based only on morphology and the final decision made by time-lapse | Can be made on the day of transfer (1 hour between primary and seconday decision).
  In the time-lapse Group we plan to compare the decision made based solely on morphology (Before the KID score is made) and after the KID score has been applied.

CONTACTS AND LOCATIONS:
Locations (11):
- Livio Reykjavik, Reykjavik, Iceland
- Livio Oslo, Oslo, Norway
- Sweden (9):
  - Livio Falun, Falun
  - Fertilitetscentrum Livio Göteborg, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Livio Malmö, Malmo
  - Karolinska Universtetssjukhuset, Stockholm
  - Livio Gärdet, Stockholm
  - Livio Kungsholmen, Stockholm
  - Sophiahemmet, Stockholm
  - Livio Umeå, Umeå

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ahlstrom A, Lundin K, Lind AK, Gunnarsson K, Westlander G, Park H, Thurin-Kjellberg A, Thorsteinsdottir SA, Einarsson S, Astrom M, Lofdahl K, Menezes J, Callender S, Nyberg C, Winerdal J, Stenfelt C, Jonassen BR, Oldereid N, Nolte L, Sundler M, Hardarson T. A double-blind randomized controlled trial investigating a time-lapse algorithm for selecting Day 5 blastocysts for transfer. Hum Reprod. 2022 Apr 1;37(4):708-717. doi: 10.1093/humrep/deac020. PMID 35143661